CLINICAL TRIAL: NCT01553097
Title: Neurocognitive Impairment in Women With Early Stage Breast Cancer
Brief Title: Examining a Common Complaint of Women Who Receive Chemotherapy for Breast Cancer- Cognitive Difficulty
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12321; 5P30NR011403 (NIH)
Record Dates: First submitted 2011-11-10; First posted 2012-03-13 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Neurocognitive Impairment; Quality of Life
Keywords: Breast Cancer; Neurocognitive Impairment; Quality of Life; Cytokines
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 cc of blood in a BD Vacutainer® tube preserved with 5.4mg K2 EDTA for the cytokine assay
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- women with stage I or II BC with adjuvant chemotherapy: women with Stage I or II BC who
  1. have undergone surgical treatment (biopsy, lumpectomy or mastectomy) and;
  2. will be receiving adjuvant chemotherapy
  Interventions: Other: Neurocognitive impairment observation
- women with Stage I or II BC without adjuvant therapy: Women with stage I or II BC who
  1. Have undergone surgical treatment (biopsy, lumpectomy or mastectomy) \
  2. will not be receiving adjuvant chemotherapy
  Interventions: Other: Neurocognitive impairment observation
- Healthy control: healthy education-age-matched women without cancer
  Interventions: Other: Neurocognitive impairment observation

INTERVENTIONS:
Other: Neurocognitive impairment observation — None - observational

SUMMARY:
This longitudinal project will investigate a common complaint of women who receive chemotherapy for breast cancer- cognitive difficulty. The relationships of fatigue, stress, and depression to cognitive difficulties will be examined. The findings should lead to interventions to decrease the effects of these problematic side effects.

DETAILED DESCRIPTION:
Most women with breast cancer are diagnosed in the early stages of the disease (Stage I and II) and 90% of these can expect to survive at least 5 years. Adjuvant chemotherapy regimens for breast cancer are often associated with complaints of cognitive changes, mostly the inability to concentrate and memory lapses that may persist in some women long after chemotherapy has ended. These changes are frequently accompanied by reports of a triad of behavioral conditions: fatigue, increased stress, and depressive symptoms. Biologically, cytokine release patterns play an important role in regulation of the immune system and normal CNS function, including neural cell repair and metabolism of neurotransmitters-both critical for normal cognitive functioning. Thus, the theoretical underpinnings of this research are embedded in the biobehavioral (mind-body) model which characterizes the multidimensional interactions among the mind, neuroendocrine, and immune systems. The purpose of this prospective, longitudinal project of 100 women is to determine whether there are differences in cognitive functioning and related behavioral conditions (fatigue, perceived stress, and depressive symptoms) in women in each of 3 groups: those with early stage BC treated with surgery and chemotherapy, women with early stage BC treated with surgery and without chemotherapy and an age-gender-education-matched healthy cohort without cancer. The primary aim of the project is to examine the relationships among fatigue, perceived stress, and depressive symptoms and neurocognitive impairment. A secondary aim is to explore the relationships among key behavioral and biological markers that may explain underlying mechanisms for development of neurocognitive impairment. In particular, this project will explore pro- and anti-inflammatory cytokine patterns and their potential associations with neurocognitive functioning. For the primary aim, the mixed linear model will be used to test for differences between the groups. For analysis of the secondary aim variable reduction stage and correlation will be used. The strength of this project is its biobehavioral approach to discerning underlying mechanisms of neurocognitive impairment in women with early stage BC receiving adjuvant chemotherapy. In addition, three other common behavioral conditions associated with BC and/or chemotherapy, fatigue, perceived stress, and depressive symptoms, will be evaluated for their potentially confounding effects on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* read and speak English
* be physically able to take the computerized test (press the keyboard space bar and numerical keys "1" and "2" without difficulty)
* have an ECOG Performance Status score < 2.154
* capable of providing informed consent.

Exclusion Criteria:

* psychiatric impairment, such as organic brain disorders, mental retardation, active psychoses or dissociative disorders, or unstable and/or severe depressive illness.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the two BC groups will be recruited from the Massey Cancer Center (MCC) clinical sites in Richmond, VA. Healthy volunteers will be recruited throughout the VCU Health System and through women's groups throughout the greater Richmond, VA area. The PI will provide physicians and clinical nurses an overview of the research and work with them to identify potential project participants. Participants will be provided oral and written information about the research and given an opportunity to ask questions or discuss the project with family or significant others.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
test neurocognitive function, using CNSVS, of the three groups while adjusting for fatigue, perceived stress, and depressive symptoms. | baseline
test for neurocognitive function, using CNSVS, of the three groups while adjusting for fatigue, perceived stress, and depressive symptoms. | 4 months
test for neurocognitive function, using CNSVS, of the three groups while adjusting for fatigue, perceived stress, and depressive symptoms. | 9 months

SECONDARY OUTCOMES:
test level of inflammatory markers in order to explore the relationships between key behavioral and biological markers that may explain underlying mechanisms for development of neurocognitive impairment (NI). | baseline, month 4 and month 9

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Grapp, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virnigia Commonwealth University, Richmond, Virginia, United States